CLINICAL TRIAL: NCT03113890
Title: McLean and Genomind Prospective Study of Pharmacogenetic Testing
Brief Title: McLean and Genomind Prospective Study
Acronym: GPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Genomind, LLC (Industry)
Responsible Party: Principal Investigator, Kerry Ressler, Principal Investigator, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017P000380
Record Dates: First submitted 2017-04-01; First posted 2017-04-14 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Major Depressive Disorder; PTSD
Keywords: pharmacogenetic testing; genomic; assay; PTSD; pharmacodynamic; pharmacokinetic; psychiatric disorders
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Mental Disorders

STUDY DESIGN:
Intervention Model Description: The investigators will enroll 200 inpatient subjects over 2 years who will donate saliva/undergo a cheek swab to collect DNA for the Genecept assay. For 100 patients in the assay-guided group (AGG), study doctors will receive the Genecept report prior to patient discharge and use it to guide psychoeducation and medication management. For the additional 100 inpatients, treating clinicians will not receive the report during the patient's inpatient stay (treatment as usual, TAU). Study Doctors will receive the assay report for patients in the treatment-as-usual group at the 3-month followup period. Thus this group will serve as the control group for the outcomes related to Genecept-guided decision making.
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assay Guided Group (AGG) (Experimental): These patients will undergo a cheek swab to collect DNA for the Genecept assay. Study doctors will receive the Genecept report prior to patient discharge and use it to guide psychoeducation and medication management.
  Interventions: Genetic: Phlebotomy - Folate; Genetic: Cheek Swab; Other: Self-report surveys
- Treatment as Usual (TAU) (Other): Thus this group will serve as the control group for the outcomes related to Genecept-guided decision making. These patients will undergo a cheek swab to collect DNA for the Genecept assay. Study doctors will receive the Genecept report at the 12-week follow up visit (12 weeks after patient discharge) and will use it to guide psychoeducation. The Study Doctors will not receive the report during the patient's inpatient stay (treatment as usual, TAU). Clinicians will receive the assay report for patients in the treatment-as-usual group at the 3-month followup period.
  Interventions: Genetic: Phlebotomy - Folate; Genetic: Cheek Swab; Other: Self-report surveys

INTERVENTIONS:
Genetic: Phlebotomy - Folate — This will be a blood draw performed at Visit 1 for Folate (one 7mL tube)
Genetic: Cheek Swab — Participants will undergo a cheek swab to then be analyzed using the Genecept Assay created by Genomind, Inc. This will occur once during Visit 1.
Other: Self-report surveys — At visit 1 and at visit 3 and 4, participants will be asked to complete self report diagnostic surveys and surveys related to the objective aims of the study.

SUMMARY:
This is a three month naturalistic prospective, randomized, open label study of pharmacogenetic testing and clinical outcomes in inpatients across diagnoses, including Treatment Resistant Depression (TRD) with or without Post-Traumatic Stress Disorder (PTSD), recruiting from the Short Term Unit at McLean Hospital.

Specifically, the investigators will enroll 200 inpatient subjects over 2 years who will donate saliva/undergo a cheek swab to collect DNA for the Genecept assay. For 100 patients in the assay-guided group, treating Clinicians will receive the Genecept report prior to patient discharge and use it to guide psychoeducation and medication management. For the additional 100 inpatients, treating clinicians will not receive the report during the patient's inpatient stay (treatment as usual. Clinicians will receive the assay report for patients in the treatment-as-usual group at the 3-month followup period. Thus this group will serve as the control group for the outcomes related to Genecept-guided decision making.

DETAILED DESCRIPTION:
Importance / Relevance:

Psychiatric disorders are etiologically complex and clinically heterogeneous which makes them challenging to diagnose and effectively treat. Thus, they pose a huge societal burden and involve substantial costs in human and financial terms. Specifically in the U.S., mental health disorders including MDD and PTSD account for 6.2% of the nation's health care spending. Major depressive disorder and schizophrenia are listed by the World Health Organization as being among the top 10 leading causes of years lost due to disability.

The primary means of treating major mental illness remains psychotropic-based, whether alone or in combination with psychotherapy. Despite an ever-growing number of medication options, however, outcomes remain significantly suboptimal. In the landmark Sequenced Treatment Alternatives to Relieve Depression (STAR*D) study, only 37% achieved remission with first-line therapy with a selective serotonin reuptake inhibitor (SSRI), whereas 16.3% withdrew completely from treatment due to drug intolerance. In the Clinical Antipsychotic Trails of Intervention Effectiveness (CATIE), over 74% eventually discontinued study medication either because of lack of efficacy or tolerability. And in the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD) trial, up to 75% patients experienced symptoms relapse over the course of follow-up.

With the advent of the genomics revolution, and precision and personalized medicine, tailoring patients' medication treatment to their individual pharmacokinetic and pharmacodynamic characteristics is being increasingly embraced by various fields of medicine. Testing is currently available for cardiovascular, cancer, autoimmune, infectious, and psychiatric illnesses, etc. In fact, over 140 US Food and Drug Administration (FDA)-approved drugs have pharmacogenomic-based guidelines; at least 27 of these are psychotropics, including Celexa for which the FDA specially recommend dose-reduction for P450 CYP2C19 poor metabolizers due to the risk of QT prolongation (FDA, 2014). Yet the vast majority of Celexa-prescribing clinicians are unaware of which of their patients are among the 3% of poor metabolizers or the 20% of the intermediate metabolizers who are also at increased risk.

Genomind, a Pennsylvania-based personalized medicine company, provides genetic testing with the Genecept™ Assay that can help clinicians optimize treatment for their patients with mental illness. This test is an alternative to the traditional trial and error approach to psychiatric drug prescribing which fails approximately 50% of the time.

The Genecept Assay identifies patient-specific genetic markers that indicate which treatments are likely to work as intended, be ineffective, or cause adverse effects. The assay is easily administered by a cheek swab test and analyzes variations in key genes that can inform treatment decisions. The assay is used to guide treatment for a broad range of psychiatric conditions including depression, anxiety, obsessive-compulsive disorder (OCD), attention deficit hyperactivity disorder (ADHD), bipolar disorder, post-traumatic stress disorder (PTSD), autism, schizophrenia, chronic pain and substance abuse. Each test provides clinicians with an easy-to-read patient report and complimentary psychopharmacogenomic consultation with Genomind's expert scientific staff (including Physicians, PhDs, and PharmDs). Additionally, the assay has been shown in peer reviewed published studies to improve patient outcomes and reduce overall medical costs.

Brief summary of procedures and recruitment:

This is a six month naturalistic prospective, randomized, open label study of pharmacogenetic testing and clinical outcomes in inpatients across diagnoses, including Treatment Resistant Depression (TRD) with or without Post-Traumatic Stress Disorder (PTSD), recruiting from the Short Term Unit at McLean Hospital.

Specifically the investigators will enroll 200 inpatient subjects over 2 years who will donate saliva/undergo a cheek swab to collect DNA for the Genecept assay. For 100 patients in the assay-guided group, treating Clinicians will receive the Genecept report prior to patient discharge and use it to guide psychoeducation and medication management. For the additional 100 inpatients, treating clinicians will not receive the report during the patient's inpatient stay (treatment as usual. Clinicians will receive the assay report for patients in the treatment-as-usual group at the 3-month followup period. Thus this group will serve as the control group for the outcomes related to Genecept-guided decision making.

Primary Objectives:

Objective 1: Does Inpatient Genetic Testing Improve Symptoms at Follow-up: This aim will test if, by the 3-month follow-up, inpatient psychopharmacogenetic testing will reduce symptoms of depression and anxiety.

Objective 2: Does Inpatient Genetic Testing Improve Readmission: This aim will test if, by the 3-month follow-up, inpatient psychopharmacogenetic testing will reduce frequency of inpatient readmission.

Secondary Objectives:

Objective 3: Does Inpatient Genetic Testing Improve Discharge Measures: This aim will test if, by discharge, inpatient psychopharmagogenetic testing enhances measures of patient satisfaction, and symptom measurement.

Objective 4: Does Inpatient Genetic Testing Improve Follow-up Measures: This aim will test if, by the time of 3-month and 6-month follow-up, inpatient psychopharmacogenetic testing will increase measures of follow-up treatment compliance, reduce time to stable medication regimen; and suicide attempts; reduce self-medication with substance of abuse.

Objective 5: Does Inpatient Genetic Testing Improve Medication Management: This aim will test, if when examined retrospectively across the discharge and 3-month data and 6-month data, inpatient psychopharmacogenetic testing will improve medication adherence, reduce number of medication trials, and reduce time-to-effective dose.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients admitted to the Short Term Unit at Mclean Ability to understand and sign informed consent. These patients cover a transdiagnostic range of severe depression, anxiety, and PTSD.
* Both genders, all ethnic backgrounds, age 18 or older
* Fluent English speakers

Exclusion Criteria:

* Involuntary hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Does Inpatient Genetic Testing Improve Symptoms at Follow-up: | 3-month follow up
  This aim will test if, by the 3-month follow-up, inpatient psychopharmacogenetic testing will reduce symptoms of depression and anxiety.
Does Inpatient Genetic Testing Improve Readmission: | 3-month follow up
  This aim will test if, by the 3-month follow-up, inpatient psychopharmacogenetic testing will reduce frequency of inpatient readmission.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry J Ressler, MD PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No